CLINICAL TRIAL: NCT05070156
Title: A Phase 1 Open-label, Single Arm Study Targeting Glypican-3 (GPC3) Chimeric Antigen Receptor Modified T Cells (CAR-T) for Treatment of Advanced Hepatocellular Carcinoma
Brief Title: B010-A Injection for Treating Patients With GPC3 Positive Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tongji University (Other)
Collaborators: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Principal Investigator, Qing Xu, Principle Investigator, Tongji University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B010-A-001
Record Dates: First submitted 2021-09-10; First posted 2021-10-07 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — Biological Products; Vaccines; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: B010-A injection for patient with GPC3 Positive Hepatocellular Carcinoma (Experimental)
  Interventions: Biological: Biological/Vaccine: Low-dose group; Biological: Biological/Vaccine: Mid-dose group; Biological: Biological/Vaccine: High-dose group

INTERVENTIONS:
Biological: Biological/Vaccine: Low-dose group — 1.0×105/kg positive CAR-T cells injection. 2-n doses will be evaluated by the investigator if participant is qualify for certain condition.
Biological: Biological/Vaccine: Mid-dose group — 2.0×105/kg positive CAR-T cells injection. 2-n doses will be evaluated by the investigator if participant is qualify for certain condition.
Biological: Biological/Vaccine: High-dose group — 3.0×105/kg positive CAR-T cells injection. 2-n doses will be evaluated by the investigator if participant is qualify for certain condition.

SUMMARY:
This is an Open-label, Single Arm study to observe the safety and tolerability of B010-A in the treatment of advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
All subjects participating in this study will receive peripheral blood mononuclear cell collection to produce B010-A injection products after enrollment. Subjects may receive bridging anti-cancer therapy while waiting for the production of B010-A injection. All subjects need to undergo baseline assessment before receiving cell infusion. For all subjects, the baseline assessment includes weight, body surface area, vital signs, physical examination, ECOG score, laboratory examination, coagulation function, etiological examination, 12-lead ECG, echocardiogram, cytokine testing, Tumor marker detection and ICE score, etc. Each subject will receive lymphodepletion prior to B010-A infusion, and dose-limiting toxicity (DLT) assessment will be performed on D28 after the first infusion.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must meet all of the following criteria to be eligible for enrollment in this study:

  1. Aged 18-75 years, male or female;
  2. Subjects with histopathologically or cytologically confirmed advanced hepatocellular carcinoma (HCC) who are ineligible for surgery or local therapy, have progressed or being intolerant to prior standard systemic therapies (systemic therapies include but are not limited to systemic chemotherapy and molecular targeted therapy), or those who have no effective treatment options at the time of enrollment as judged by the investigator;
  3. Subjects with at least one stable and evaluable intrahepatic or extrahepatic target lesion (longest diameter of non-nodal lesions ≥ 10 mm, or short axis of lymph node lesions ≥ 15 mm) at enrollment as per RECIST V1.1 criteria;
  4. Subjects with GPC3 positive (> grade 2) tumor tissue samples (> 25% tumor cells positive staining) as tested by immunohistochemistry (IHC);
  5. Subjects with Barcelona Clinic Liver Cancer Stage C (BCLC-C) hepatocellular carcinoma, or subjects with BCLC Stage B hepatocellular carcinoma who are not amenable to local therapy or have progressed after local therapy;
  6. Subjects with expected survival > 12 weeks;
  7. Subjects with liver cirrhosis of Child-Pugh grade A (5-6 points);
  8. Subjects with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
  9. Subjects with inactive hepatitis B (if HBsAg or HBcAb is positive, then HBV-DNA must be < 20 IU/mL, and HBsAg-positive patients should have been treated with antiviral therapies as per the Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2019 Edition));
  10. The largest diameter of intrahepatic tumors is < 10 cm, and the number of multiple tumors is < 10 (if pulmonary metastatic lesions are present, the number of metastatic lesions is < 6);
  11. Subjects with a venous access for mononuclear cell collection;
  12. Subjects with adequate bone marrow function that allows for lympho-depleting pre-conditioning and without contraindications for the pre-conditioning as assessed by the investigator;
  13. Subjects with liver, kidney, respiratory, cardiovascular functions, and corresponding hematological levels as defined below:

      1. Alanine aminotransferase (ALT) ≤ 5.0 × ULN, aspartate aminotransferase (AST) ≤ 5.0 × ULN, and total bilirubin ≤ 2.5 × ULN at screening;
      2. Requirements for blood coagulation at screening: prothrombin time (PT) prolongation ≤ 4 s, fibrinogen ≥ 1 g/L, activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;
      3. Serum creatinine ≤ 1.5 × ULN or endogenous creatinine clearance > 50 mL/min (Cockcroft-Gault formula) at screening;
      4. Pulmonary function at screening: finger oxygen saturation ≥ 95% at screening and prior to apheresis;
      5. Cardiac function at screening: left ventricular ejection fraction (LVEF) ≥ 50% as assessed by echocardiography within 1 month;
      6. Subjects with white blood cell count ≥ 3.0×109/L and lymphocyte count ≥ 0.5×109/L at screening (except for those receiving bridging chemotherapy), platelet count ≥ 75×109/L, hemoglobin ≥ 90 g/L, and neutrophil count ≥ 1.5×109/L (this criterion should also be met within 24 hours prior to apheresis).
  14. Female subjects of childbearing potential (all women physiologically capable of becoming pregnant) must have a negative serum pregnancy test both at screening and within 14 days prior to the first dose and are willing to use reliable contraception methods during the study (within 24 months after the first dose of cell infusion). For male subjects whose partners are women of childbearing potential, the subjects should have been surgically sterilized or agree to use reliable contraception methods during the study as well as for additional 1 year after receiving the last study treatment;
  15. Subjects with ability to understand and sign the Informed Consent Form.

Exclusion Criteria:

* Subjects who meet any of the following criteria cannot participate in this study:

  1. Having other uncured malignancies (except cervical carcinoma in situ and basal cell carcinoma of skin) within the past 5 years or at present, or hepatocellular carcinoma with brain metastases;
  2. With a history of any of the following cardiovascular diseases within the past 6 months: New York Heart Association (NYHA) Grade III or IV heart failure, cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant heart diseases, or poorly controlled high blood pressure (systolic blood pressure > 150 mm Hg, or diastolic blood pressure > 90 mm Hg), or hypotension that requires treatment with vasopressors;
  3. With metastases to the central nervous system (CNS) and clinically significant CNS disorders; with prior or clinically significant CNS diseases at screening, such as epilepsy, seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, brain organic syndrome or psychiatric disorder;
  4. With prior hepatic encephalopathy or at present;
  5. With a history of serious lung diseases, including pulmonary embolism, chronic obstructive pulmonary disease, interstitial lung disease and clinically significant abnormal findings in pulmonary function tests;
  6. With an active infection (uncontrolled active infections caused by bacteria, viruses, or fungus requiring systemic therapy) at screening, or has an unexplained fever of ≥ 38.0 °C during screening or prior to the first dose;
  7. With known active autoimmune diseases requiring immunosuppressive therapy, including biologics;
  8. With a history of organ transplantation or awaiting organ transplantation (including liver transplantation);
  9. With ≥ 50% of liver replaced by tumor, or with the main portal vein tumor thrombus, or the mesenteric vein/inferior vena cava has been invaded by tumor thrombus;
  10. With a co-infection of HBV and HCV viruses or infections caused by more than two viruses;
  11. Positive HCV-RNA, HIV antibody, or syphilis serology, or any other uncontrollable active infections;
  12. Requiring long-term antiplatelet therapy (aspirin > 300 mg/day; clopidogrel > 75 mg/day);
  13. Have received prior cell-based therapies such as targeted GPC3 therapy, TCR-T therapy, CAR-T therapy;
  14. With moderate or higher amount of pleural effusion/ascites with clinical symptoms, or have undergone drainage of pleural effusion/ascites within the past month (except for those with only small amounts of pleural effusion/ascites revealed by imaging examinations but without symptoms);
  15. With active bleeding or coagulation test abnormalities, bleeding tendency or undergoing thrombolytic, anticoagulant, or antiplatelet therapy (except those requiring heparin due to PICC or deep vein catheterization), or massive bleeding/blood loss (greater than 450 mL) within 28 days;
  16. With a history of gastrointestinal bleeding within 3 months or definite tendency of gastrointestinal bleeding (e.g., known locally active ulcer lesions, fecal occult blood positive);
  17. Having received any of the following treatments:

      1. Have received supportive care such as blood transfusion, platelet transfusion, cell growth factors (except recombinant erythropoietin) within 2 weeks prior to apheresis:
      2. Have received anti-PD-1/PD-L1 monoclonal antibody treatment within 4 weeks prior to apheresis;
      3. Have used any study drug within 4 weeks prior to apheresis, except those who have failed to respond to the study treatment or have experienced disease progression during study treatment and at least 3 half-lives have passed prior to peripheral blood mononuclear cell collection);
      4. Have undergone any surgical treatment, interventional therapy, chemoradiotherapy, ablation, targeted therapy, treatments with invasive investigational medical devices, or are receiving immunomodulatory therapy for the disease under study within 2 weeks prior to apheresis;
      5. With prior use of prednisone at doses ≥ 15 mg /day (or equivalent glucocorticoids) systemically within 2 weeks prior to apheresis, or may require long-term glucocorticoid therapy during study treatment as judged by the investigator (except those who have recently or are currently using inhaled or topical glucocorticoids);
      6. Have received any Chinese herbal medicine or Chinese patent medicine to control liver cancer within 2 weeks prior to apheresis.
  18. With previous allergic reactions to immunotherapy, have received related drugs (such as tocilizumab, cyclophosphamide), or excipients or matrix components contained in B010-A for Injection (e.g., albumin, dimethyl sulfoxide, etc.);
  19. Toxicities caused by prior treatments have not recovered to CTCAE Grade ≤ 1, except for alopecia and other events judged as tolerable by the investigator;
  20. Unable or unwilling to comply with protocol requirements as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate incidence of treatment-emergent adverse events [Safety and Tolerability] after B010-A injection. | Up to 24 months post B010-A injection.

SECONDARY OUTCOMES:
Evaluate the cellular kinetics of subjects after B010-A injection. | Up to 24 months post B010-A injection.
  Copy number of transgenes of GPC3-CAR-T (qPCR).
Evaluate the cellular kinetics of subjects after B010-A injection. | Up to 24 months post B010-A injection.
  Copy number of CAR-T cell transgene level detection (flow cytometry).
Evaluate the pharmacodynamics of subjects after B010-A injection. | Up to 24 months post B010-A injection.
  Measurement of cytokine.
Evaluate the pharmacodynamics of subjects after B010-A injection. | Up to 24 months post B010-A injection.
  Measurement of C-reactive protein (CRP).
Evaluate the preliminary efficacy of B010-A after injection. | Up to 24 months post B010-A injection.
  Measurement of free GPC3 protein in peripheral blood, and lymphocyte subpopulation.
Progression-free survival (PFS) | Up to 24 months post B010-A injection.
  Determination of the progression-free survival of all subjects
Overall survival (OS) | Up to 24 months post B010-A injection.
  Determination of the overall survival of all subjects
Objective remission rate (ORR) | Up to 24 months post B010-A injection.
  Determination of the objective remission rate of all subjects
Disease control rate (DCR) | Up to 24 months post B010-A injection.
  Determination of the disease control rate of all subjects
Duration of remission (DOR) | Up to 24 months post B010-A injection.
  Determination of the duration of remission of all subjects
Disease control Time (DDC) | Up to 24 months post B010-A injection.
  Determination of the disease control time of all subjects

CONTACTS AND LOCATIONS:
Overall Officials: Qing Xu, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China